CLINICAL TRIAL: NCT07086001
Title: Does it Work? Examining the Acceptability and Effectiveness of a Self-Directed, Web-Based Resource for Stress and Coping in University: Randomized Controlled Trial
Brief Title: Examining the Acceptability and Effectiveness of a Self-Directed, Web-Based Resource for Stress and Coping in University: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Nancy Heath, Distinguished James McGill Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-10-040; 253619 (Other Grant/Funding Number: McGill's Regional Bicentennial Campaign)
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Stress; Coping; Coping Behavior; Well-Being (Psychological Flourishing); Digital Intervention
Keywords: stress; coping; university students; digital intervention
MeSH Terms: interventions — Coping Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Directed (Experimental): Website presenting a collection of stress-management, motivation, healthy coping, well-being, and socializing resources + brief screener directing students to tailored resources based on responses to the screener (demonstrating low, moderate, or high need for support around stress and coping).
  Interventions: Behavioral: stress management and coping
- Non-directed (Experimental): Website presenting a collection of stress-management, motivation, healthy coping, well-being, and socializing resources (no tailored resource or screener was received for this group).
  Interventions: Behavioral: stress management and coping
- Waitlist Comparison (No Intervention): Did not have access to the strategies during the project, the full web-based resource was shared with the comparison group at the end of data collection.

INTERVENTIONS:
Behavioral: stress management and coping — Online intervention focusing on stress and coping in university students. All resources were grouped in five main categories: Managing Stress, Enhancing Performance, Adulting, Socialising, and Well-being. The resource was hosted on a website and presented information in several multimedia formats (i.e., text, audio, video, interactive infographic) to account for diversity of preferences. All students in the intervention groups were provided with unlimited access to the intervention. Furthermore, all students were asked to complete screener questions on their stress and coping but only students in the directed group were directed to one of three unique pages on the website based on their responses on the screening questionnaire demonstrating low, moderate, or high need for support around stress and coping.
  Arms: Directed; Non-directed

SUMMARY:
University students consistently report high levels of stress and psychological distress and identify these as key factors that negatively impact their academic performance and engagement with their studies. Supporting students in effectively coping with stress and distress is of critical importance to facilitate learning and development in university environments. To that end, technology-based approaches to delivering stress-management and well-being supports to university students have proliferated on campuses as supplemental means of supporting student stress management, coping capacity, and well-being. Indeed, online resources for students' self-directed use such as websites, apps, or on-demand workshops, are increasingly popular given their benefits in improving access to support as well as the potential for reaching students who may be reluctant to seek other forms of mental health support or are on waiting lists for more specialized services. In addition, the provision of resources for addressing stress and enhancing coping capacity is aligned with the recently proposed health theory of coping which calls for enhancing the availability of evidence-based healthy coping strategies. However, investigation into the acceptability, and even more critically the effectiveness of online, self-directed resources for non-clinical stress-management and healthy coping support is limited. Thus, this study sought to explore the acceptability and effectiveness of a self-directed, web-based resource for enhancing students' stress-management and coping capacity. Furthermore, the study also examined if there would be any added benefit of screening students to assess stress and coping needs and then directing them to specific resources to match their needs for stress-management and healthy coping support.

DETAILED DESCRIPTION:
University students' mental health and well-being have been a growing concern within higher education research and practice for many decades. For those pursuing a university education, this time in their lives often corresponds with their developmental transition to adulthood. Coined in research literature as emerging adulthood, this developmental period is distinct from adulthood conceptually and as a subjective experience. Emerging adulthood is a challenging yet unique time of exploration and settling into adult roles, often characterized as a time of feeling in-between. The transitional nature of this developmental period has implications for university students' mental health and well-being, as it is also a time where high rates of engagement in risky and unhealthy coping behaviours have been observed. Taken together, there is a clear need to enhance access to evidence-based strategies and tools to support students in effectively managing stress and enhancing their capacity to cope with distress.

To date, efforts aimed at improving student mental health and well-being in university settings have included a wide variety of interventions targeting stress, depression, anxiety, resilience, and general mental health and well-being. Increasingly, technology-based and online tools (e.g., websites, apps, chat-bots, on-demand programming) are used with several systematic and meta-analytic reviews emphasizing the promise of the technology-based approach for improving key outcomes. Self-directed or self-administered online resources have the potential to serve as supplementary support for students and offer several advantages. First, they have the potential to reach those who may not access face-to-face services, who may not meet clinical criteria for specialized treatments or are on waitlists for services, thus broadening access to evidence-based strategies and supports. Second, the self-guided format is supportive of student autonomy and confidentiality as individuals can choose when, where, and how to access information and make use of resources most aligned with their individual needs. Lastly, the online presentation of information and evidence-based strategies and techniques allows for a cost-effective, low-intensity, and adaptable (i.e., possibility to update and/or change based on contextual needs) means to supplement existing mental health and well-being services on campus.

Despite the advantages described above and emerging evidence of effectiveness for using online, self-directed approaches to student support, research examining the effectiveness and acceptability of this approach is in its infancy. In addition, it is unclear to what extent online, self-directed programming and resources are integrated into the university setting and utilized beyond their initial effectiveness trials. Notably, even when interventions and programs for student mental health and well-being are shown to be effective, they are often only shared with students through the universities' health and wellness center, relying on students to proactively seek help to access these services. This poses a challenge because research consistently shows that university students exhibit low levels of help-seeking, leading to the underutilization of many services and resources despite a high demand. Thus, there is an urgent need to explore alternative approaches for resource delivery that facilitate students' universal and ongoing access to self-directed support options to comprehensively address stress and coping needs.

In summary, despite the rapid proliferation of online self-guided resources for university students, research examining the effectiveness of this approach for improving stress and coping is still in its infancy. Further research is needed to address gaps and deepen our understanding of what works best and how in the area of supporting university students' stress-management and coping capacity. Thus, using a randomized-controlled design, this study sought to examine the acceptability and effectiveness of a web-based, self-directed resource for university students containing evidence-based strategies for stress-management and healthy coping. In addition, this study examined whether there would be any added benefit of using a screening approach to direct students to personalized resources aligned with their identified needs. Participants were randomly assigned to one of three groups; directed to personalized resources aligned with needs, non-directed but received all resources, and waitlist comparison. Main outcomes assessed were participant ratings of acceptability, stress, coping (coping self-efficacy and coping behaviours), and well-being over time.

Specifically, the first objective (1) was to examine potential group differences (directed and non-directed resource groups only) in students' acceptability of the web-based resource over time. It was hypothesized that (H1) acceptability would be higher in the directed group when compared to the non-directed over time. The second objective (2) was to examine the effectiveness of the online self-directed resources in terms of group differences (directed, non-directed, comparison) on outcome measures (i.e., stress, coping, and well-being) and in terms of differences in scores over time between baseline, post, and follow-up measures. It is hypothesized (H2a) that the directed group will show stronger improvements across stress, coping, and well-being outcomes over time than both the non-directed group and the comparison group. It is also hypothesized (H2b) that the non-directed group will show significant improvements across study outcomes relative to the comparison group. Lastly, the third objective (3) was to examine the effectiveness of the overall web-based, self-directed resource in terms of group differences (resource group; merged directed and non-directed versus the comparison group) on outcome measures and in terms of change in scores over time between baseline, post, and follow-up measures (i.e., stress, coping, and well-being). It is hypothesized (H3) that the resource group will show significant improvements across study outcomes in relation to the comparison group.

Participants who expressed interest in participating in the study were asked to complete a brief online demographics survey to facilitate their random assignment into the three different conditions within the study; namely, directed to resources based on reported need in the screening questionnaire (Group 1: directed), non-directed sharing of all resources (Group 2: non-directed), and waitlist comparison (Group 3: comparison). Responses to the demographic questionnaire were used to ensure comparable samples across the different conditions in terms of participants' age, gender, and program of study. Following random assignment to the different conditions, all participants were asked to complete the baseline measures and the screening questionnaire (described in the measures section below). Although all participants were asked to complete the brief screening questionnaire, only those in the directed group subsequently received personalized instruction on how to use the resources and strategies provided in the online resource.

Group 1 (Directed) Immediately following the completion of the baseline survey, Group 1 were given access to the website presenting a collection of stress-management, motivation, healthy coping, well-being, and socializing resources. Additionally, based on their answers to the brief screener, Group 1 were directed to one of three unique pages on the website based on their responses on the screening questionnaire demonstrating low, moderate, or high need for support around stress and coping. The directing process was automated using a scoring algorithm within the survey platform used in this study (i.e., Qualtrics).

Group 2 (Non-directed) Participants in Group 2 followed the same procedure as Group 1; however, they did not receive any personalized instruction and were simply directed to the home page of the website containing resources.

Group 3 (Comparison) Participants in Group 3 constituted the waitlist comparison group. As such, they did not have access to any of the strategies hosted on the website during the data collection phase of the study. Participants in Group 3 were asked to complete online surveys identical to those completed by Groups 1 and 2. Although Group 3 did not have access to the strategies during the project, the full web-based resource was shared with the comparison group at the end of data collection.

In terms of data collection timeline, all groups completed measures regarding their stress, coping, and well-being at the start of the study (Baseline: T1), four weeks after the start of the study (Post: T2), and eight weeks following the start of the study (Follow-up: T3). In addition, participants in Groups 1 and 2 completed a brief check-in to assess resource acceptability two weeks after baseline which is when the resources were initially shared with participants.

ELIGIBILITY:
Inclusion Criteria:

* University student

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Change in Stress | Week 1, 5 & 9
  The Perceived Stress Scale (PSS; Cohen, 1988) is a widely used self-report measure of individuals' perception of stress. This measure contains 10 items in which participants indicate their experience of stress on a 5-point Likert scale (0 = never to 4 = very often). Items were adapted to reflect experiences during the past week and include statements such as "In the past week, how often have you felt difficulties were piling up so high that you could not overcome them?" Ratings were averaged across items such that higher scores represented greater perceived stress. The PSS has good reliability (Cronbach's α = .89), construct validity, and predictive validity with reports of psychological and physical symptoms.

SECONDARY OUTCOMES:
Acceptability of the Resource | Week 1, 5 & 9
  A researcher-developed measure aligned with the Kirkpatrick New World Model for program evaluation. Specifically, a total of 11 items assessed participants' (1) overall satisfaction with the resource (8 items; e.g., "I found the website useful for me"; "The strategies presented in the website helped me better understand how to manage my stress and improve my wellness"; "I found that the website presented valuable strategies and techniques" rated on a 4-point Likert scale; 1= strongly disagree to 4= strongly agree), (2) frequency of actual and planned use of strategies (2 item; i.e., "Over the past two weeks, how often did you use the strategies presented on the website?" and "Over the coming weeks, how often do you plan to use the strategies presented on the website?" Rated on a 4-point Likert scale; 1 = every day to 4= never) as well as (3) a single item to rate perceived impact for their well-being (i.e., "Over the past two weeks, how would you rate the impact of the strategie
Change in Coping Self-efficacy | Week 1, 5 & 9
  The Coping Self-Efficacy Scale (CSES; Chesney et al., 2006) which is a measure of one's confidence in effectively engaging in coping behaviors in the face of challenges. This measure contains 26 items in which participants indicate confidence in their coping strategies when it comes to handling challenges and stressors on an 11-point Likert scale (0 = cannot do at all to 10 = certain can do). The CSES states, "When things aren't going well for you, or when you're having problems, how confident or certain are you that you can do the following:" and include statements such as "find solutions to your most difficult problems" and "see things from the other person's point of view during a heated argument." Higher scores on the CSES represent higher coping-self efficacy.
Change in Coping Behaviours | Week 1, 5 & 9
  The Coping Index (CI) was used to assess students' engagement in healthy and unhealthy coping behaviours over the duration of the study. The CI is a 20-item measure of engagement with healthy (10 items) and unhealthy (10 items) coping behaviours which are aligned with the health theory of coping framework (Stallman, 2020). Participants are asked to indicate how often they engage in each behaviour listed when they feel stressed or distressed on a 4-point Likert scale (0= I don't do this at all to 3= I do this most of the time). Higher scores on the healthy coping subscale indicate greater frequency of engagement in healthy coping behaviours, and higher scores on the unhealthy coping subscale indicate greater frequency of engagement in unhealthy coping in response to stress or distress. This measure has been found to have satisfactory test-retest reliability in previous studies (α = .71) (Stallman, 2019).
Change in Well-being | Week 1, 5 & 9
  The Warwick-Edinburg Mental Well-Being Scale (WEMWBS; Tennant et al., 2007), which is a measure of positive mental health and consists of 14 positively worded items. Participants are asked to rate statements such as "I've been feeling good about yourself" on a 5-point Likert scale according to their experience over the past 2 weeks (1= none of the time; 5= all of the time). The WEMWBS has demonstrated good internal consistency in student (α = .89) and general population samples (α = .91) and was found to be psychometrically robust in validation studies (Stewart-Brown et al., 2011; Tennant et al., 2007).

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma L, Zhang Y, Cui Z. Mindfulness-based interventions for prevention of depressive symptoms in university students: A meta-analytic review. Mindfulness. 2019;10:2209-2224. doi:10.1007/s12671-019-01192-w
- [Background] Ang WHD, Lau ST, Cheng LJ, Chew HSJ, Tan JH, Shorey S, et al. Effectiveness of resilience interventions for higher education students: A meta-analysis and metaregression. Journal of Educational Psychology. 2022;114(7):1670-1694. doi:10.1037/edu0000719
- [Background] Conley CS, Durlak JA, Kirsch AC. A Meta-analysis of universal mental health prevention programs for higher education students. Prev Sci. 2015 May;16(4):487-507. doi: 10.1007/s11121-015-0543-1. PMID 25744536
- [Background] Böke BN, Mills DJ, Mettler J, Heath NL. Stress and coping patterns of university students. Journal of College Student Development. 2019;60(1):85-103. doi:10.1353/csd.2019.0005
- [Background] Swanson JA. Trends in literature about emerging adulthood: Review of empirical studies. Emerging Adulthood. 2016;4(6):391-402. doi:10.1177/2167696816630468
- [Background] Arnett JJ. Emerging adulthood. A theory of development from the late teens through the twenties. Am Psychol. 2000 May;55(5):469-80. PMID 10842426
- [Background] Conley CS, Kirsch AC, Dickson DA, Bryant FB. Negotiating the transition to college: Developmental trajectories and gender differences in psychological functioning, cognitive-affective strategies, and social well-being. Emerging Adulthood. 2014;2(3):195-210. doi:10.1177%2F2167696814521808
- [Background] Hill M, Farrelly N, Clarke C, Cannon M. Student mental health and well-being: Overview and Future Directions. Ir J Psychol Med. 2024 Jun;41(2):259-266. doi: 10.1017/ipm.2020.110. Epub 2020 Nov 27. PMID 33243317
- [Background] Stallman HM. Health theory of coping. Australian Psychologist. 2020;55(4) :295-306. doi :10.1111/ap.12465
- [Background] Harrer M, Adam SH, Fleischmann RJ, Baumeister H, Auerbach R, Bruffaerts R, Cuijpers P, Kessler RC, Berking M, Lehr D, Ebert DD. Effectiveness of an Internet- and App-Based Intervention for College Students With Elevated Stress: Randomized Controlled Trial. J Med Internet Res. 2018 Apr 23;20(4):e136. doi: 10.2196/jmir.9293. PMID 29685870
- [Background] Stallman HM. Psychological distress in university students: A comparison with general population data. Australian Psychologist. 2010;45(4):249-257. doi:10.1080/00050067.2010.482109
- [Background] Lattie EG, Adkins EC, Winquist N, Stiles-Shields C, Wafford QE, Graham AK. Digital Mental Health Interventions for Depression, Anxiety, and Enhancement of Psychological Well-Being Among College Students: Systematic Review. J Med Internet Res. 2019 Jul 22;21(7):e12869. doi: 10.2196/12869. PMID 31333198
- [Background] Sharp J, Theiler S. A review of psychological distress among university students: Pervasiveness, implications and potential points of intervention. International Journal for the Advancement of Counselling. 2018;40:193-212. doi:10.1007/s10447-018-9321-7